CLINICAL TRIAL: NCT02876458
Title: EMERGEncy Versus Delayed Coronary Angiogram in Survivors of Out-of-hospital Cardiac Arrest With no Obvious Non Cardiac Cause of Arrest
Brief Title: EMERGEncy Versus Delayed Coronary Angiogram in Survivors of Out-of-hospital Cardiac Arrest
Acronym: EMERGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150914; 2016-A00413-48 (Other: ANSM); PHRC-15-15-0570 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2016-07-31; First posted 2016-08-23 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Coronary angiogram; Survival rate; Neurological sequel
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate coronary angiogram (Other): An immediate coronary angiogram will be performed
  Interventions: Other: Immediate coronary angiogram
- Delayed coronary angiogram (Other): A delayed coronary angiogram (between 48 to 96 hours) will be performed
  Interventions: Other: Delayed coronary angiogram

INTERVENTIONS:
Other: Immediate coronary angiogram — An immediate coronary angiogram will be performed
  Arms: Immediate coronary angiogram
Other: Delayed coronary angiogram — A delayed coronary angiogram (between 48 to 96 hours) will be performed
  Arms: Delayed coronary angiogram

SUMMARY:
Sudden cardiac death (SCD) remains a major public health issue with a low survival rate. The most common cause of SCD is acute coronary artery occlusion. Several registry based studies suggest that coronary angiography (CA) performed at admission followed if necessary by coronary angioplasty improves in-hospital and long term survival. Recent guidelines recommend performing an immediate CA in all survivors of SCD with no obvious non cardiac cause of arrest. However there is a lack of randomized data on this topic.

Several retrospective studies have shown that if the post-resuscitation electrocardiogram (ECG) shows ST segment elevation, the probability of finding an acute coronary artery lesion during the CA is high (70-80%). In contrast, if no ST segment elevation is present the probability is low (15-20%).

Performing an immediate CA in all survivors of SCD can be challenging. It requires admitting these patients to centers with an intensive care unit and facilities allowing 24/24 7/7 CA. It may increase the delay of performing other therapeutic modalities such as CT brain or thorax scan to determine the cause of SCD. Performing the CA 48 to 96 hours after admission would facilitate the management of these difficult patients. However if the cause of the arrest is a coronary artery occlusion and there is a delay in reperfusion, the rate of post-arrest shock and the mortality may increase. Therefore a randomized study comparing immediate versus delayed (between 48 to 96 hours) CA in survivors of SCD with no obvious non-cardiac cause of arrest is warranted.

DETAILED DESCRIPTION:
The design consists in a multicenter national randomized open parallel group trial.

All eligible patients with SCD will be included and randomized by the Emergency Medical Service (EMS) to one of the 2 following arms: immediate CA vs delayed CA. Patients randomized in the immediate CA group will be admitted directly to the catheterization laboratory. Patients randomized in the delayed CA will be admitted to the intensive care unit and a CA will be planned 48 to 96 hours after admission. Investigators can perform the CA in the delayed group < 48 hours if the following events appear:

* ST segment elevation or new left bundle branch block on the ECG
* Shock unresponsive to inotropes
* "Electrical storm" (repeated Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF))
* Segmental hypokinesia or akinesia on an echocardiogram

Echocardiography and assessment of neurological status are done at discharge form the Intensive Care Unit, at hospital discharge and during the follow-up visits (90 and 180 days).

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital SCD with return of spontaneous circulation
* Age ≥ 18 years of age
* No obvious non-cardiac cause of arrest
* Admitted to a center with an intensive care unit and a 24 hours a day, 7 days a week interventional cardiology department
* Affiliation to the French Social Security Health Care plan

Exclusion Criteria:

* Age < 18 years of age
* In-hospital SCD
* No return of spontaneous circulation
* Presence of ST segment elevation
* Suspected non-cardiac aetiology (trauma, respiratory, neurological, etc.)
* Presence of co-morbidities with life expectancy of less than a year
* Pregnancy
* Adults subject to a legal protection measure (guardianship or tutelage measure)
* Participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Survival with no or minimal neurological sequel | 180 days
  Survival rate with no or minimal neurological sequel (CPC (cerebral performance category) 1 or 2) at 6 months after inclusion

SECONDARY OUTCOMES:
Shock | 48 hours
  The rate of shock during the first 48 hours between immediate and delayed CA
Arrhythmia | 48 hours
  The rate of VT/VF during the first 48 hours between immediate and delayed CA
The evolution of left ventricular ejection fraction evolution | 180 days
  Changes in left ventricular ejection fraction between baseline and 180 days assessed by echocardiogram between immediate and delayed CA
CPC score | 180 days
  The rate of neurological sequel assessed by the CPC score between immediate and delayed CA
Glasgow Outcome Scale Extended score (GOSE) | 180 days
  The rate of neurological sequel assessed by the GOSE between immediate and delayed CA
Overall survival rate | 180 days
  The overall survival rate between immediate and delayed CA
Hospital stay length | 180 days
  The length of hospital stay between immediate and delayed CA

CONTACTS AND LOCATIONS:
Overall Officials: Christian Spaulding, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- European Georges Pompidou Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauw-Berlemont C, Lamhaut L, Diehl JL, Andreotti C, Varenne O, Leroux P, Lascarrou JB, Guerin P, Loeb T, Roupie E, Daubin C, Beygui F, Boissier F, Marjanovic N, Christiaens L, Vilfaillot A, Glippa S, Prat JD, Chatellier G, Cariou A, Spaulding C; EMERGE Investigators. Emergency vs Delayed Coronary Angiogram in Survivors of Out-of-Hospital Cardiac Arrest: Results of the Randomized, Multicentric EMERGE Trial. JAMA Cardiol. 2022 Jul 1;7(7):700-707. doi: 10.1001/jamacardio.2022.1416. PMID 35675081